CLINICAL TRIAL: NCT00496561
Title: Evaluation of Early Clinical and Immunological Efficacy of Specific Immunotherapy to Dust Mites in Children With Asthma
Brief Title: Effect of Specific Immunotherapy to Dust Mites in Children With Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Professor, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNN-149-06-KE
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: asthma; immunotherapy; children; regulatory T cells; ECP; PC20M; Quality of Life; Symptoms score; Spirometry
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): subcutaneous immunotherapy (House Dust Mites)
  Interventions: Biological: subcutaneous immunotherapy (House Dust Mites)
- 2 (Placebo Comparator): placebo of subcutaneous immunotherapy (House Dust Mites)
  Interventions: Other: placebo of subcutaneous immunotherapy (House Dust Mites)

INTERVENTIONS:
Biological: subcutaneous immunotherapy (House Dust Mites) — subcutaneous immunotherapy (House Dust Mites)
  Arms: 1
Other: placebo of subcutaneous immunotherapy (House Dust Mites) — placebo of subcutaneous immunotherapy (House Dust Mites)
  Arms: 2

SUMMARY:
The aim of the study is to assess the effect of specific immunotherapy (SIT) to dust mites on clinical symptoms, reliever drugs usage, inhaled glucocorticosteroid usage, quality of life, lung function, chosen markers of inflammation, induction of regulatory lymphocytes, bronchial hyperreactivity with methacholine, and presence and type of allergy after two years of SIT in children with asthma.

DETAILED DESCRIPTION:
Specific immunotherapy is the only one causal treatment method of atopic diseases including bronchial asthma in children.

The aim of the study is to assess the effect of specific immunotherapy (SIT) to dust mites on clinical symptoms,reliever drugs usage, inhaled glucocorticosteroid usage, quality of life, lung function, chosen markers of inflammation, induction of regulatory lymphocytes, bronchial hyperreactivity with methacholine, and presence and type of allergy after two years of SIT in children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* patients allergic to house dust mites
* patients with moderate bronchial asthma
* patients with controlled asthma
* patients who were qualified for immunotherapy and gave written informed consent for immunotherapy (active treatment group)
* patients who were qualified for immunotherapy and did not agree with this kind of treatment - did not give written informed consent for immunotherapy (control group)

Exclusion Criteria:

* patients allergic for other perennial and seasonal allergens
* patients with other chronic diseases that either put the patient at risk when participating in the study or could influence the results of the study or the patient's ability to participate in the study as judged by the investigator
* medications that resulted in patient exclusion included:anti-parasites or oral corticosteroids within 6 months before the first visit.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-08; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
clinical symptoms, reliever drugs usage, controller medication usage, quality of life, lung function, chosen markers of inflammation (ECP, specific IgE, specific IgG) induction of regulatory lymphocytes (Treg) - Foxp3 mRNA expression | baseline (first visit), after 3 months (second visit), 12 months (third visit), 24 months (fourth visit)

SECONDARY OUTCOMES:
bronchial hyperreactivity with methacholine, and presence and type of allergy after two years of SIT (skin prick tests) | after 24 months from first visit (fourth visit)

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Stelmach, MD, PhD, Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Dorota Jurałowicz, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, Lodz, Poland